CLINICAL TRIAL: NCT00652756
Title: Evaluation of the Versamed iVent in the Transport of Patients Receiving Mechanical Ventilation
Acronym: iVent
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequately
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7299; 000
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Respiration, Artificial
Keywords: Respiration, Artificial; Transportation of Patients; Intubation, Intratracheal; Tracheostomy
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patient is placed on a transport ventilator.
  Interventions: Device: Use of ventilator during patient transport (Versamed iVent)
- 2 (Other): Patient is ventilated using the current standard at this institution.
  Interventions: Other: Bag-valve ventilation

INTERVENTIONS:
Device: Use of ventilator during patient transport (Versamed iVent) — The goal of the transport ventilator is to provide optimal ventilation.
  Other Names: Versamed iVent ventilator
  Arms: 1
Other: Bag-valve ventilation — Use of bag-valve ventilation during patient transport.
  Other Names: Use of manual resuscitator during transport.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the use of the VersaMed iVent ventilator in the acute care setting, hypothesizing that, in comparison to the standard approach, the use of the VersaMed will facilitate transport and reduce transport-associated complications while providing equivalent ventilatory support and transport success rates for both intubated patients and patients receiving noninvasive ventilation.

DETAILED DESCRIPTION:
Transporting acute-care patients who require mechanical ventilation within a hospital can be fraught with hazards. Prior studies have revealed a high level of transport-associated complications including episodes of hypertension, hypoxemia, respiratory arrest, and death (1). In many institutions, the preferred method of transporting intubated patients is to use manual ventilation with a resuscitator bag, an approach that fully occupies one member of the transport team. Using a transport ventilator involves taking an intubated patient who has been placed on one ventilator and switching the patient to the transport ventilator; until now, transport ventilators had not been designed to match the capabilities of the more robustly engineered critical care ventilators.

The use of noninvasive ventilation (NIV) to treat patients with COPD exacerbations and other forms of respiratory failure has increased because of its demonstrated efficacy in reducing the need for intubation as well as morbidity and mortality (2). None of the ventilators usually used for noninvasive ventilation was designed for in-patient transport.

Currently, the standard of care in this institution is to transport intubated patients receiving mechanical ventilation by using a manual resuscitation bag and to transport patients receiving NIV by placing the patient on oxygen therapy without ventilatory support.

The VersaMed iVent ventilator was designed to treat respiratory failure in the acute care setting. The device is suitable for patients who are intubated as well as for patients receiving noninvasive ventilation, has a backup battery so that it can function during transport, and has been approved by the FDA for invasive and noninvasive mechanical ventilation. This device permits continuity of mechanical ventilation virtually regardless of patient status.

We propose to evaluate the utility of the VersaMed iVent ventilator in the acute care setting, hypothesizing that, in comparison to the standard approach, the use of the VersaMed will facilitate transport, reduce transport-associated complications, and provide equivalent ventilatory support and transport-success rates for both intubated patients and patients receiving NIV.

References

1. Braman SS, Dunn SM, Amico CA, Millman RP. Complications of intrahospital transport in critically ill patients. Ann Intern Med 1987; 107:469-73.
2. Mehta S, Hill NS. Noninvasive ventilation-state of the art. Am J Respir Crit Care Med 2001; Feb; 163(2):540-77.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the trial will be receiving mechanical ventilation in the emergency department, critical care, and other patient care areas; and will require transport within the hospital.

Exclusion Criteria:

* Patient must be at least eighteen years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To determine whether using a ventilator during patient transport has better outcomes than the current approach to transport. | One year (estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S. Hill, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States